CLINICAL TRIAL: NCT03547908
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Fixed Dose Combination of Bictegravir/Emtricitabine/Tenofovir Alafenamide Versus Dolutegravir + Emtricitabine/Tenofovir Disoproxil Fumarate in Treatment Naïve, HIV-1 and Hepatitis B Co-Infected Adults
Brief Title: Safety and Efficacy of Bictegravir/Emtricitabine/Tenofovir Alafenamide Versus Dolutegravir + Emtricitabine/Tenofovir Disoproxil Fumarate in Treatment Naive, HIV-1 and Hepatitis B Co-Infected Adults
Acronym: Alliance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-380-4458; 2018-000926-79 (EudraCT Number)
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: HIV-1/HBV Co-Infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Blinded Phase: B/F/TAF (Experimental): Participants who are HIV-1 and HBV co-infected and treatment-naïve will receive Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) fixed-dose combination (FDC) tablet in addition to placebo to match (PTM) dolutegravir (DTG) tablet and PTM FDC emtricitabine/ tenofovir desoproxil fumarate (F/TDF) tablet for 96 weeks.
  Interventions: Drug: B/F/TAF; Drug: Placebo to match DTG; Drug: Placebo to match F/TDF
- Blinded Phase: DTG+F/TDF (Active Comparator): Participants who are HIV-1 and HBV co-infected and treatment-naïve will receive DTG and FDC F/TDF in addition to PTM B/F/TAF for 96 weeks.
  Interventions: Drug: DTG; Drug: F/TDF; Drug: Placebo to match B/F/TAF
- Open-label Extension Phase: B/F/TAF from B/F/TAF (Experimental): After Week 96, participants will continue to take their blinded study drug and attend visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants in a country where B/F/TAF FDC is not available will be given the option to receive B/F/TAF FDC in an open-label extension phase for up to 48 weeks, or until the product becomes accessible through an access program, or until Gilead elects to discontinue the study in that country, whichever occurs first.
  Interventions: Drug: B/F/TAF
- Open-label Extension Phase: B/F/TAF from DTG+F/TDF (Experimental): After Week 96, participants will continue to take their blinded study drug and attend visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants in a country where B/F/TAF FDC is not available will be given the option to receive B/F/TAF FDC in an open-label extension phase for up to 48 weeks, or until the product becomes accessible through an access program, or until Gilead elects to discontinue the study in that country, whichever occurs first.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: B/F/TAF — 50/200/25 mg B/F/TAF FDC tablet administered orally once daily, without regard to food
  Other Names: Biktarvy®
  Arms: Blinded Phase: B/F/TAF; Open-label Extension Phase: B/F/TAF from B/F/TAF; Open-label Extension Phase: B/F/TAF from DTG+F/TDF
Drug: Placebo to match DTG — Tablet administered orally once daily, without regard to food
  Arms: Blinded Phase: B/F/TAF
Drug: Placebo to match F/TDF — Tablet administered orally once daily, without regard to food
  Arms: Blinded Phase: B/F/TAF
Drug: DTG — 50 mg tablet administered orally once daily, without regard to food
  Arms: Blinded Phase: DTG+F/TDF
Drug: F/TDF — 200/300 mg tablet administered orally once daily, without regard to food
  Other Names: Truvada®
  Arms: Blinded Phase: DTG+F/TDF
Drug: Placebo to match B/F/TAF — Tablet administered orally once daily, without regard to food
  Arms: Blinded Phase: DTG+F/TDF

SUMMARY:
The primary objective of this study is to evaluate the efficacy of fixed-dose combination (FDC) of bictegravir/emtricitabine/ tenofovir alafenamide (B/F/TAF) versus dolutegravir (DTG) + emtricitabine/tenofovir disoproxil fumarate (F/TDF) in treatment-naïve and HIV-1 and hepatitis B virus (HBV) adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Human immunodeficiency virus type 1 (HIV-1) co-infection:

  * Must be HIV antiretroviral treatment naive with plasma HIV-1 ribonucleic acid (RNA) ≥ 500 copies/mL at screening
  * ≤ 10 days of prior therapy with any antiretroviral agent, including lamivudine and entecavir, following a diagnosis of HIV-1 infection (except the use for pre-exposure prophylaxis (PrEP) or post-exposure prophylaxis (PEP), up to one month prior to screening)
  * Screening genotype report must show sensitivity to emtricitabine (FTC) and tenofovir (TFV). This report will be provided by Gilead Sciences. Alternatively, if genotype results from a local laboratory obtained ≤ 90 days prior to screening visit date show sensitivity to these drugs, this genotype will be acceptable to fulfill this inclusion criterion in the event that the genotype obtained at screening is not yet available and all other inclusion/exclusion criteria have been confirmed
* HBV co-infection:

  * Must be hepatitis B virus (HBV) treatment naive (defined as < 12 weeks of oral antiviral treatment)
  * Screening HBV deoxyribonucleic acid (DNA) ≥ 2000 IU/mL
* Hepatic transaminases (aspartate aminotransferase (AST) and alanine aminotransferase (ALT)) ≤ 10 x upper limit of normal (ULN)
* Total bilirubin ≤ 2.5 x ULN

Key Exclusion Criteria:

* Hepatitis C virus (HCV) antibody positive and HCV RNA detectable
* Individuals experiencing decompensated cirrhosis (eg, ascites, encephalopathy, or variceal bleeding) or with Child-Pugh-Turcotte (CPT) C impairment
* Current alcohol or substance use judged by the Investigator to potentially interfere with study compliance
* Active, serious infections (other than HIV-1 and HBV infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Day 1
* Participation in any other clinical trial, including observational studies, without prior approval from the sponsor is prohibited while participating in this trial

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (69):
- United States (4):
  - Midway Immunology & Research, Ft. Pierce, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Be Well Medical Center, Berkley, Michigan
  - The Crofoot Research Center, INC (DBA: Gordon E. Crofoot MD PA), Houston, Texas
- China (10):
  - Beijing Ditan Hospital Capital Medical University, Beijing
  - Beijing YouAn Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing
  - The First Hospital of Changsha, Changsha
  - Chengdu Public Health Clinical Center, Chengdu
  - Guangzhou Eighth people's Hospital, Guangzhou
  - 1st Affiliated Hospital of Zhejiang University, Hangzhou
  - The Second Hospital of Nanjing, Nanjing
  - Shanghai Public Health Clinical Center, Shanghai
  - Third People's Hospital Of Shenzhen, Shenzhen
- Instituto Dominicano de Estudios Virologicos (IDEV), Santo Domingo, Dominican Republic
- Hôpital de la Croix Rousse, Lyon, France
- Greece (4):
  - Evaggelismos General Hospital of Athens, Athens
  - Korgialenio-Benakio Greek Red Cross General Hospital, Athens
  - Laiko General Hospital, Athens
  - AHEPA University Hospital of Thessaloniki, Thessaloniki
- Hong Kong (3):
  - Prince of Wales Hospital, Hong Kong
  - Queen Elizabeth Hospital (QEH), Hong Kong
  - Princess Margaret Hospital, Kowloon
- Japan (8):
  - National Hospital Organization Nagoya Medical Center, Aichi
  - University of the Ryukyus Hospital, Okinawa
  - Osaka City General Hospital, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - The Jikei University Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
  - Yokohama City University Hospital, Yokohama
- Malaysia (9):
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Raja Perempuan Zainab II, Kota Bharu
  - Queen Elizabeth Hospital, Kota Kinabalu
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu
  - Sarawak General Hospital, Kuching
  - Hospital Pulau Pinang, Pulau Pinang
  - Sungai Buloh Hospital, Sungai Buloh
- Hope Clinical Research, San Juan, Puerto Rico
- South Korea (2):
  - Pusan National University Hospital, Busan
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (8):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Santa Lucia, Cartagena
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital de Canarias, Santa Cruz de Tenerife
  - Hospital General Universitario de Valencia, Valencia
  - CHUVI - Hospital Universitario Alvaro Cunqueiro, Vigo
- Taiwan (9):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei City Hospital Linsen, Chinese Medicine and Kunming Branch, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Ministry of Health and Welfare Taoyuan General Hospital, Taoyuan
- Thailand (7):
  - Thai Red Cross AIDS Research Centre (HIV-NAT), Bangkok
  - Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok
  - Siriraj Hospital, Bangkok
  - Faculty of Medicine, Chiang Mai University, Chiang Mai
  - Chiang Rai Reginal Hospital, Chiang Rai
  - Srinagarind Hospital, Khon Kaen
  - Bamrasnaradura Infectious Diseases Institute, Nonthaburi
- Turkey (Türkiye) (2):
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Background] Avihingsanon, A. 2022. Week 48 results of a Phase 3 randomized controlled trial of bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) vs dolutegravir + emtricitabine/tenofovir Disoproxil Fumarate (DTG+F/TDF) as initial treatment in HIV/HBV-coinfected adults (ALLIANCE). AIDS, 29 July 29-2 August 2022, Montréal, Québec, Canada.
- [Background] Avihingsanon A, Lu H, Leong CL, Hung CC, Koenig E, Kiertiburanakul S, Lee MP, Supparatpinyo K, Zhang F, Rahman S, D'Antoni ML, Wang H, Hindman JT, Martin H, Baeten JM, Li T; ALLIANCE Study Team. Bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir, emtricitabine, and tenofovir disoproxil fumarate for initial treatment of HIV-1 and hepatitis B coinfection (ALLIANCE): a double-blind, multicentre, randomised controlled, phase 3 non-inferiority trial. Lancet HIV. 2023 Oct;10(10):e640-e652. doi: 10.1016/S2352-3018(23)00151-0. Epub 2023 Jul 23. PMID 37494942
- [Background] D'Antoni ML, Andreatta K, Chang S, Cox S, Hindman JT, Avihingsanon A, Martin H, VanderVeen LA, Callebaut C. Brief Report: HIV-1 Resistance Analysis of Participants With HIV-1 and Hepatitis B Initiating Therapy With Bictegravir/Emtricitabine/Tenofovir Alafenamide or Dolutegravir Plus Emtricitabine/Tenofovir Disoproxil Fumarate: A Subanalysis of ALLIANCE Data. J Acquir Immune Defic Syndr. 2024 Aug 1;96(4):380-384. doi: 10.1097/QAI.0000000000003434. Epub 2024 Jun 21. PMID 40788226
- [Background] Avihingsanon A, Lu H, Leong CL, Hung C-C, Kiertiburanakul S, Lee M-P, Supparatpinyo K, Zhang F, Hindman JT, Wang H, Liu H and Li T. Factors Associated with HBV Response to B/F/TAF vs. DTG + F/TDF at W96 in People with HIV-1 and HBV. CROI, March 3-6, 2024.
- [Background] Avihingsanon A, Lu H, Leong C, Hung C, Koenig E, Kiertiburanakul S, et al. Week-96 results of ALLIANCE, a Phase 3, randomized, double-blind study comparing bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) versus dolutegravir + emtricitabine/tenofovir disoproxil fumarate (DTG+F/TDF) in treatment-naive people with both HIV-1 and hepatitis B. 12th International AIDS Society Conference on HIV Science 2023, 23-26 July.
- [Background] D'Antoni M, Andreatta K, Cox S, Chang S, Hindman J, Martin H, et al. HIV-1 resistance analysis of treatment-naive participants with HIV-1 and hepatitis B coinfection receiving bictegravir/emtricitabine/tenofovir alafenamide or dolutegravir + emtricitabine/tenofovir disoproxil fumarate. European Meeting on HIV and Hepatitis 2023, 7-9 June, Rome, Italy.
- [Background] Avihingsanon A, Leong C, Hung C, Koenig E, Lee M, Supparatpinyo K, et al. Predictors of hepatitis B treatment response in people with HIV-1/HBV coinfection. Conference on Retroviruses and Opportunistic Infections (CROI) 2023, 19-22 February; Seattle, Washington.
- [Background] Avihingsanon A, Lu H, Leong C, Hung C, Koenig E, Kiertiburanakul S, et al. Week 48 results of a Phase 3 randomized controlled trial of bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) vs dolutegravir + emtricitabine/tenofovir disoproxil fumarate (DTG+F/TDF) as initial treatment in HIV/HBV coinfected adults (ALLIANCE). AIDS (Conference) 2022, 29 July 2 August; Montréal, Québec, Canada.
- [Derived] D'Antoni ML, Boopathy AV, Andreatta K, Chang S, Hindman JT, Avihingsanon A, VanderVeen LA, Callebaut C. Brief Report: HIV-1 Resistance Analysis of Participants With HIV-1 and Hepatitis B Receiving Bictegravir/Emtricitabine/Tenofovir Alafenamide or Dolutegravir Plus Emtricitabine/Tenofovir Disoproxil Fumarate Through the Open-Label Extension of the ALLIANCE Study. J Acquir Immune Defic Syndr. 2025 Dec 1;100(4):342-346. doi: 10.1097/QAI.0000000000003749. PMID 40857111
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-380-4458

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the North American, Asian, and European regions.
Pre-assignment Details: 381 participants were screened.
Groups:
- Blinded Phase: B/F/TAF: Participants who were HIV-1 and HBV co-infected and treatment-naïve received Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) fixed-dose combination (FDC) tablet orally, once daily without regard to food for 96 weeks. Participants also received placebo to match (PTM) dolutegravir (DTG) tablet and PTM FDC emtricitabine/ tenofovir desoproxil fumarate (F/TDF) tablet orally once daily without regard to food for 96 weeks.
- Blinded Phase: DTG + F/TDF: Participants who were HIV-1 and HBV co-infected and treatment-naïve received DTG (50 mg) tablet + F/TDF (200/300 mg) FDC tablet, orally, once daily without regard to food for 96 weeks. Participants also received PTM FDC B/F/TAF tablet, orally, once daily without regard to food for 96 weeks.
- Open-Label Extension Phase: B/F/TAF From B/F/TAF; Open-Label Extension Phase: B/F/TAF From DTG+F/TDF: After Week 96, participants continued their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, if safety and efficacy of B/F/TAF FDC was demonstrated for the HIV-1 and HBV coinfected participants, in a country where B/F/TAF FDC was not available, participants were given the option to receive 48 weeks of open-label B/F/TAF until the product became accessible through an access program, or until Gilead elected to discontinue the study in that country, whichever occurred first.
Period: Blinded Phase
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF | Open-Label Extension Phase: B/F/TAF From B/F/TAF | Open-Label Extension Phase: B/F/TAF From DTG+F/TDF
Started | 122 | 122 | 0 | 0
Completed | 111 | 113 | 0 | 0
Not Completed | 11 | 9 | 0 | 0
Not completed — Lost to Follow-up | 3 | 3 | 0 | 0
Not completed — Withdrew Consent | 2 | 3 | 0 | 0
Not completed — Investigator's Discretion | 2 | 1 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0
Not completed — Non-compliance With Study Drug | 0 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Randomized But Never Treated | 1 | 0 | 0 | 0
Period: Open-label Extension Phase
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF | Open-Label Extension Phase: B/F/TAF From B/F/TAF | Open-Label Extension Phase: B/F/TAF From DTG+F/TDF
Started | 0 | 0 | 95 (Out of 111 participants who completed the Blinded Phase, 95 entered the Open-label Extension Phase.) | 89 (Out of 113 participants who completed the Blinded Phase, 89 entered the Open-label Extension Phase.)
Completed | 0 | 0 | 91 | 88
Not Completed | 0 | 0 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safely Analysis Set included participants who were randomized into the study and received at least 1 dose of study drug.
Groups:
- Blinded Phase: B/F/TAF: Participants who were HIV-1 and HBV coinfected and treatment-naïve received Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) fixed-dose combination (FDC) tablet orally, once daily without regard to food for 96 weeks. Participants also received placebo to match (PTM) dolutegravir (DTG) tablet and PTM FDC emtricitabine/ tenofovir desoproxil fumarate (F/TDF) tablet orally once daily without regard to food for 96 weeks.
- Blinded Phase: DTG + F/TDF: Participants who were HIV-1 and HBV coinfected and treatment-naïve received DTG (50 mg) tablet + F/TDF (200/300 mg) FDC tablet, orally, once daily without regard to food for 96 weeks. Participants also received PTM FDC B/F/TAF tablet, orally, once daily without regard to food for 96 weeks.
- Total: Total of all reporting groups
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF | Total
Number analyzed (Participants) | 121 | 122 | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 120 | 121 | 241
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (9.2) | 33 (9.4) | 33 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 112 | 120 | 232
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 17
  Not Hispanic or Latino | 114 | 112 | 226
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 108 | 106 | 214
  Race: White | 10 | 9 | 19
  Race: Black | 2 | 6 | 8
  Race: Other | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 55 | 39 | 94
  China | 27 | 29 | 56
  Malaysia | 15 | 22 | 37
  Taiwan | 5 | 7 | 12
  Dominican Republic | 4 | 6 | 10
  Turkey | 4 | 5 | 9
  Japan | 2 | 5 | 7
  Spain | 4 | 3 | 7
  Hong Kong | 2 | 3 | 5
  United States | 1 | 2 | 3
  South Korea | 2 | 0 | 2
  Puerto Rico | 0 | 1 | 1
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 282 (193.1) | 266 (194.3) | 274 (193.5)
CD4 Percentage [Mean (Standard Deviation); unit: percentage of CD4 cells] | 16.0 (8.62) | 14.8 (8.25) | 15.4 (8.44)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm (Co-primary Endpoint)
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. Percentages were rounded-off.
Time Frame: Week 48
Population: The Full Analysis Set included all participants who were randomized into the study, received at least 1 dose of study drug, and had at least 1 postbaseline HIV-1 RNA or HBV DNA result while on study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF
Number analyzed (Participants) | 119 | 122
percentage of participants | 95.0 | 91.0
Statistical Analysis 1: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Non-Inferiority — A sample size of 240 participants randomized in a 1:1 ratio to 2 treatment groups, achieved 90% power to detect a non-inferiority margin of 12% between the 2 treatment groups. For the sample size and power computation, it is assumed that both treatment groups have a response rate of 91% (based on Gilead Studies GS-US-380-1489 and GS-US-380-1490), that the non-inferiority margin is 12%, and that the significance level of the test is at a one-sided 0.025 level; Difference in Percentages = 4.1, 95.001% CI 2-sided [-2.5 to 10.8] — The difference in percentages of participants between groups and their 95.001% confidence intervals (CI)s were calculated based on Mantel-Haenszel (MH) proportions adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL)
Statistical Analysis 2: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Superiority; p = 0.2113, Cochran-Mantel-Haenszel; The p-value was calculated from Cochran-Mantel-Haenszel (CMH) test stratified by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL)

2. Primary Outcome: Percentage of Participants With Plasma Hepatitis B Virus (HBV) DNA < 29 IU/mL at Week 48 as Defined by Missing = Failure Approach (Co-primary Endpoint)
Description: This outcome measure was analyzed using a Missing = Failure approach. In this approach, all missing data were treated as HBV DNA ≥ 29 IU/mL. Percentages were rounded-off.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF
Number analyzed (Participants) | 119 | 122
percentage of participants | 63.0 | 43.4
Statistical Analysis 1: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Non-Inferiority — A sample size of 240 participants provided 81% power to detect a non-inferiority margin of 12% between the 2 treatment groups. This assumed that both treatment groups have a response rate of 88% (based on Gilead Studies GS-US-320-0108 and GS-US-320-0110), that the non-inferiority margin is 12%, and that the significance level of the test is at a one-sided 0.025 level; Difference in Percentages = 16.6, 95.001% CI 2-sided [5.9 to 27.3]; The difference in percentages of participants with HBV DNA < 29 IU/mL between treatment groups and its 95.001% CI were calculated based on the MH proportions adjusted by baseline HBeAg status (positive vs negative) and baseline HBV DNA category (< 8 log10 IU/mL vs ≥ 8 log10 IU/mL)
Statistical Analysis 2: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Superiority; p = 0.0023, Cochran-Mantel-Haenszel; The p-value was from CMH test stratified by baseline HBeAg status (positive vs negative) and HBV DNA category (< 8 log10 IU/mL vs ≥ 8 log10 IU/mL)

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which was defined as a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. Percentages were rounded-off.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF
Number analyzed (Participants) | 119 | 122
percentage of participants | 87.4 | 87.7
Statistical Analysis 1: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Superiority; p = 0.9427, Cochran-Mantel-Haenszel — P-value for the superiority test comparing the percentages of participants with HIV-1 RNA < 50 copies/mL between treatment groups was from the CMH test stratified by baseline HIV-1 RNA stratum (≤ 100,000 vs > 100,000 copies/mL); Difference in Percentages = -0.3, 95% CI 2-sided [-8.9 to 8.3] — The difference in percentages of participants with HIV-1 RNA < 50 copies/mL between treatment groups and its 95% CI were calculated based on the MH proportions adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs > 100,000 copies/mL)

4. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF
Number analyzed (Participants) | 117 | 116
cells/µL | 200 (139.3) | 175 (124.7)
Statistical Analysis 1: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Other; p = 0.1701, ANOVA; The p-value was calculated using ANOVA model adjusted by the baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL); Difference in least squares mean (LSM) = 24, 95% CI 2-sided [-10 to 58] — The difference in least squares means and its 95% CI were calculated using ANOVA model adjusted by the baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL)

5. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 96
Time Frame: Baseline, Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF
Number analyzed (Participants) | 109 | 113
cells/uL | 261 (161.6) | 229 (174.0)
Statistical Analysis 1: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Other; p = 0.1853, ANOVA — P-value was from ANOVA model adjusted by the baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in Least Squares Means = 30, 95% CI 2-sided [-14 to 74] — Difference in least squares means (Diff in LSM), and its 95% CI were from ANOVA model adjusted by the baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL)

6. Secondary Outcome: Change From Baseline in Percentage of CD4 Cells at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4 cells
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF
Number analyzed (Participants) | 117 | 116
percentage of CD4 cells | 8.43 (4.1) | 7.75 (4.3)
Statistical Analysis 1: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Other; p = 0.2839, ANOVA; [statistical method as in outcome 4, analysis 1]; Difference in least squares mean (LSM) = 0.59, 95% CI 2-sided [-0.49 to 1.67] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Change From Baseline in Percentage of CD4 Cells at Week 96
Time Frame: Baseline, Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4 cells
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF
Number analyzed (Participants) | 108 | 112
percentage of CD4 cells | 10.69 (5.047) | 10.42 (5.096)
Statistical Analysis 1: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Other; p = 0.8456, ANOVA — P-value was from ANOVA model adjusted by the baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in LSM = 0.13, 95% CI 2-sided [-1.20 to 1.46] — Difference in LSM and its 95% CI were from ANOVA model adjusted by the baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL)

8. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 29 IU/mL at Week 96
Description: as for outcome 2
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF
Number analyzed (Participants) | 119 | 122
percentage of participants | 74.8 | 70.5
Statistical Analysis 1: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; The difference in percentages of participants with HBV DNA < 29 IU/mL between treatment groups and its 95% CI were calculated based on the MH proportions adjusted by baseline HBeAg status (positive vs negative) and baseline HBV DNA category (< 8 log10 IU/mL vs ≥ 8 log10 IU/mL); Test type: Superiority — P-value for the superiority test comparing the percentages of participants with HBV DNA < 29 IU/mL between treatment groups was from the CMH test stratified by baseline HBeAg status (positive vs negative) and baseline HBV DNA category (< 8 log10 IU/mL vs ≥ 8 log10 IU/mL); p = 0.6367, Cochran-Mantel-Haenszel; Difference in Percentages = 2.6, 95% CI 2-sided [-8.3 to 13.4]

9. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) Normalization at Week 48 by American Association for the Study of Liver Diseases (AASLD) Criteria
Description: ALT normalization was defined as an ALT value that changed from above the normal range at baseline to within the normal range at the given post baseline visit. The upper limit of the normal range (ULN) for ALT using the 2018 AASLD normal range was ≤ 25 U/L for females and ≤ 35 U/L for males. The Missing = Failure approach was used for this analysis. Percentages were rounded off.
Time Frame: Week 48
Population: Participants in the Full Analysis Set with Baseline ALT > ULN were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF
Number analyzed (Participants) | 60 | 47
percentage of participants | 73.3 | 55.3
Statistical Analysis 1: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Other; p = 0.0655, Cochran-Mantel-Haenszel; P-value was calculated from CMH tests stratified by baseline HBeAg status (positive vs negative) and HBV DNA (< 8 log10 IU/mL vs ≥ 8 log10 IU/mL); Difference in Percentages = 17.1, 95% CI 2-sided [-1.5 to 35.7] — The difference in percentages of participants between groups and their 95% CIs were calculated based on MH proportions adjusted by baseline HBeAg status (positive vs negative) and baseline HBV DNA (< 8 log10 IU/mL vs ≥ 8 log10 IU/mL)

10. Secondary Outcome: Percentage of Participants With ALT Normalization at Week 96
Description: ALT normalization was defined as an ALT value that changed from above the normal range at baseline to within the normal range at the given post baseline visit. The upper limit of the normal range (ULN) for ALT using the 2018 AASLD normal range was ≤ 25 U/L for females and ≤ 35 U/L for males. The Missing = Failure approach was used for this analysis. Percentages were rounded-off.
Time Frame: Week 96
Population: Participants in the Full Analysis Set with Baseline ALT > ULN were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF
Number analyzed (Participants) | 60 | 47
percentage of participants | 71.7 | 57.4
Statistical Analysis 1: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Other; p = 0.1253, Cochran-Mantel-Haenszel; P-value was from the CMH tests stratified by baseline HBeAg status (positive vs negative) and baseline HBV DNA (< 8 log10 IU/mL vs >= 8 log10 IU/mL); Difference in Percentages = 14.1, 95% CI 2-sided [-4.3 to 32.6] — Difference in the proportion between treatment groups and its 95% CI were calculated based on the MH proportions adjusted by baseline HBeAg status (positive vs negative) and baseline HBV DNA (< 8 log10 IU/mL vs >= 8 log10 IU/mL)

11. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at Week 48
Description: HBsAg loss was defined as qualitative HBsAg changing from positive at baseline to negative at a post baseline visit. HBsAg seroconversion was defined as HBsAg loss and HBsAb changes from negative or missing at baseline to positive at a post baseline visit. The Missing = Failure approach was used for this analysis. Percentages were rounded-off.
Time Frame: Week 48
Population: The Serologically Evaluable Full Analysis Set for HBsAg loss/seroconversion included all participants who were in the Full Analysis Set and with HBsAg positive and HBsAb negative or missing at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF
Number analyzed (Participants) | 119 | 121
percentage of participants | 12.6 | 5.8
Statistical Analysis 1: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Other; p = 0.0591, Cochran-Mantel-Haenszel; P-value was from the CMH tests stratified by baseline HBeAg status (positive vs negative)and baseline HBV DNA (< 8 log10 IU/mL vs ≥ 8 log10 IU/mL); Difference in Percentages = 7.1, 95% CI 2-sided [-0.8 to 15.0] — Difference in the percentages between treatment groups and its 95% CI were calculated based on the MH proportions adjusted by baseline HBeAg status (positive vs negative) and baseline HBV DNA (< 8 log10 IU/mL vs ≥ 8 log10 IU/mL)

12. Secondary Outcome: Percentage of Participants With HBsAg Loss at Week 96
Description: as for outcome 11
Time Frame: Week 96
Population: Participants in the Serologically Evaluable Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF
Number analyzed (Participants) | 119 | 121
percentage of participants | 22.7 | 14.0
Statistical Analysis 1: Comparison: Blinded Phase: B/F/TAF vs Blinded Phase: DTG + F/TDF; Test type: Other; p = 0.0655, Cochran-Mantel-Haenszel — P value was from the CMH test stratified by baseline HBeAg status (positive vs negative) and baseline HBV DNA (< 8 log10 IU/mL vs ≥ 8 log10 IU/mL). Statistically significant values are shown in bold; Difference in Percentages = 9.3, 95% CI 2-sided [-0.7 to 19.2] — Differences in percentages between treatment groups and their 95% CI were calculated based on MH proportions adjusted by baseline HBeAg status (positive vs negative) and baseline HBV DNA (< 8 log10 IU/mL vs ≥ 8 log10 IU/mL)

ADVERSE EVENTS:
Time Frame: Adverse Events: Up to the last dose date plus 30 days (maximum exposure: 5.1 years); All-Cause Mortality: Up to 5.3 years
Description: All-Cause Mortality: All Randomized Analysis Set included all participants who were randomized into the study.
  Adverse Events: The Safely Analysis Set included participants who were randomized into the study and received at least 1 dose of study drug.
Groups:
- Blinded Phase: B/F/TAF: Participants who were HIV-1 and HBV coinfected and treatment-naïve received Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) fixed-dose combination (FDC) tablet orally, once daily without regard to food for 96 weeks. Participants also received placebo to match (PTM) dolutegravir (DTG) tablet and PTM emtricitabine/ tenofovir desoproxil fumarate (F/TDF) tablet orally once daily without regard to food for 96 weeks.
- Blinded Phase: DTG + F/TDF: Participants who were HIV-1 and HBV coinfected and treatment-naïve received DTG (50 mg) tablet + F/TDF (200/300 mg) FDC tablet, orally, once daily without regard to food for 96 weeks. Participants also received PTM B/F/TAF tablet, orally, once daily without regard to food for 96 weeks.
- Open-Label Extension Phase: B/F/TAF From B/F/TAF; Open-Label Extension Phase: B/F/TAF From DTG+F/TDF: After Week 96, participants continued their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, if safety and efficacy of B/F/TAF FDC was demonstrated for the HIV-1 and HBV coinfected participants, in a country where B/F/TAF FDC was not available, participants were given the option to receive open-label B/F/TAF until the product became accessible through an access program, or until Gilead elected to discontinue the study in that country, whichever occurred first.
Arm/Group | Blinded Phase: B/F/TAF | Blinded Phase: DTG + F/TDF | Open-Label Extension Phase: B/F/TAF From B/F/TAF | Open-Label Extension Phase: B/F/TAF From DTG+F/TDF
All-Cause Mortality (participants affected / at risk) | 2/122 | 1/122 | 1/95 | 0/89
Serious Adverse Events (participants affected / at risk) | 17/121 | 16/122 | 4/95 | 2/89
Other Adverse Events (participants affected / at risk) | 102/121 | 98/122 | 42/95 | 40/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Phase: B/F/TAF (N=121) | Blinded Phase: DTG + F/TDF (N=122) | Open-Label Extension Phase: B/F/TAF From B/F/TAF (N=95) | Open-Label Extension Phase: B/F/TAF From DTG+F/TDF (N=89)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Rhegmatogenous retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Death, not otherwise specified (General disorders) | 1 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 3 | 6 | 0 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 1 | 0 | 0
Dengue haemorrhagic fever (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 1
Hepatic amoebiasis (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Mycotoxicosis (Infections and infestations) | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Alcoholic seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Phase: B/F/TAF (N=121) | Blinded Phase: DTG + F/TDF (N=122) | Open-Label Extension Phase: B/F/TAF From B/F/TAF (N=95) | Open-Label Extension Phase: B/F/TAF From DTG+F/TDF (N=89)
Diarrhoea (Gastrointestinal disorders) | 13 | 11 | 2 | 6
Gastritis (Gastrointestinal disorders) | 8 | 2 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 7 | 2 | 1 | 0
Influenza like illness (General disorders) | 7 | 2 | 1 | 1
Pyrexia (General disorders) | 17 | 16 | 1 | 3
Acute hepatitis C (Infections and infestations) | 9 | 2 | 0 | 0
Covid-19 (Infections and infestations) | 48 | 52 | 5 | 4
Folliculitis (Infections and infestations) | 1 | 7 | 0 | 0
Latent syphilis (Infections and infestations) | 7 | 6 | 5 | 1
Nasopharyngitis (Infections and infestations) | 18 | 10 | 7 | 5
Secondary syphilis (Infections and infestations) | 7 | 7 | 1 | 1
Syphilis (Infections and infestations) | 8 | 11 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 22 | 20 | 7 | 7
Vaccination complication (Injury, poisoning and procedural complications) | 5 | 7 | 0 | 0
Alanine aminotransferase increased (Investigations) | 12 | 15 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 7 | 10 | 1 | 1
Weight increased (Investigations) | 13 | 12 | 6 | 6
Abnormal weight gain (Metabolism and nutrition disorders) | 4 | 3 | 3 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | 6 | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 9 | 1 | 0
Dizziness (Nervous system disorders) | 5 | 10 | 1 | 1
Headache (Nervous system disorders) | 13 | 9 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 10 | 9 | 2 | 0
Hypertension (Vascular disorders) | 8 | 4 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT03547908/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan - Interim Analysis (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT03547908/SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan - Final Analysis (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT03547908/SAP_002.pdf